CLINICAL TRIAL: NCT07294352
Title: Comparison of Intrathecal Nalbuphine Versus Intrathecal Tramadol as Adjuvants in Subarachnoid Block for Lower Limb Orthopaedic Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Principal Investigator, Khadija Zubair, Dr. Khadija Zubair, CMH Lahore Medical College and Institute of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 566/2024
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Adjuvants, Anesthesia; Subarachnoid Block
Keywords: Subarachnoid block; Adjuvants
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tramadol group (Active Comparator): Intrathecal tramadol 20mg + bupivacaine 0.5%
  Interventions: Drug: Intrathecal tramadol with spinal anesthsia
- Intrathecal nalbuphine (Experimental): Intrathecal nalbuphine 1 mg + bupivacaine 0.5%
  Interventions: Drug: Intrathecal nalbuphine and spinal anesthesia

INTERVENTIONS:
Drug: Intrathecal tramadol with spinal anesthsia — intrathecal tramadol 20mg with Hyperbaric 0.5% bupivacaine
  Arms: Tramadol group
Drug: Intrathecal nalbuphine and spinal anesthesia — intrathecal nalbuphine 1mg with 0.5% Hyperbaric Bupivacaine
  Arms: Intrathecal nalbuphine

SUMMARY:
This study compares the use of intrathecal nalbuphine versus intrathecal tramadol as adjuvant agents to local anaesthetics in subarachnoid block for lower-limb orthopaedic surgeries. The primary objective is to determine whether there is a meaningful difference between the two drugs in terms of quality and duration of intraoperative and postoperative analgesia. Secondary outcomes include onset and efficacy of sensory and motor block, time to first rescue analgesia, incidence of adverse effects, and perioperative hemodynamic stability. By evaluating these parameters, the study aims to identify which adjuvant provides superior analgesic benefits with fewer side effects in patients undergoing lower-limb orthopedic procedures.

DETAILED DESCRIPTION:
The effectiveness of Intrathecal Nalbuphine 1mg versus Intrathecal Tramadol 20mg as adjuvant to 0.5% hyperbaric bupivacaine in Subarachnoid block for orthopaedic surgeries of the lower limbs is studied. Primary outcomes of the study are onset of sensory block, onset of motor block, intraoperative hemodynamic stability and postoperative analgesia measured on visual analog scale. Secondary outcomes were incidence of side-effects and the need for rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1 and 2 Undergoing surgical correction of lower limb fracture

Exclusion Criteria:

* hypersensitivity to opioids or local anesthetics patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Duration of spinal anesthesia | up to 24 hours post operatively
  Time until first rescue analgesia at VAS <4. (Visual Analog scale measures subjective pain intensity on a continuous scale. Score 0 means no pain while 10 means most pain possible)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharma A, Chaudhary S, Kumar M, Kapoor R. Comparison of nalbuphine versus fentanyl as intrathecal adjuvant to bupivacaine for orthopedic surgeries: A randomized controlled double-blind trial. J Anaesthesiol Clin Pharmacol. 2021 Oct-Dec;37(4):529-536. doi: 10.4103/joacp.JOACP_270_18. Epub 2022 Jan 6. PMID 35340949